CLINICAL TRIAL: NCT02065765
Title: An International Single-Arm Protocol to Provide Expanded Access to Ramucirumab for the Treatment of Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Following Disease Progression After Prior Fluoropyrimidine and/or Platinum-Containing Chemotherapy
Brief Title: International Expanded Access Program to Provide Ramucirumab for the Treatment of Metastatic Gastric Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 14945; I4T-MC-JVCP (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Gastric Cancer; Metastatic Adenocarcinoma of the Gastroesophageal Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab

INTERVENTIONS:
Biological: Ramucirumab — Administered intravenously (IV)
  Other Names: LY3009806; IMC-1121B

SUMMARY:
The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the compassionate use program.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed gastric carcinoma, including gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma. (Participants with adenocarcinoma of the distal esophagus are eligible if the primary tumor involves the GEJ)
* The participant has metastatic disease or locally recurrent, unresectable disease
* The participant has measureable or evaluable disease as determined by standard computed tomography (CT) or magnetic resonance imaging (MRI) imaging. Examples of evaluable, nonmeasurable disease include gastric, peritoneal, or mesenteric thickening in areas of known disease, or peritoneal nodules that are too small to be considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* The participant has experienced disease progression during treatment or within 4 months after the last dose of first-line therapy for metastatic disease, or during treatment, or within 6 months after the last dose of adjuvant therapy

  o Acceptable prior chemotherapy regimens for this protocol are combination chemotherapy regimens that include platinum and/or fluoropyrimidine components. Regimens including a third agent, such as an anthracycline or a taxane, are acceptable provided a fluoropyrimidine and/or a platinum were used.
* The participant has resolution to Grade ≤1 (or to Grade ≤2 in the case of neuropathy) by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (with the exception of alopecia)
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1
* The participant has adequate hepatic function
* The participant does not have:

  * cirrhosis at a level of Child-Pugh B (or worse) or
  * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* The participant has adequate renal function as defined by a serum creatinine ≤1.5 times the upper limit of normal (ULN), or creatinine clearance (measured via 24-hour urine collection) ≥40 milliliter per minute (mL/minute)
* The participant's urinary protein is ≤1+ on dipstick or routine urinalysis (UA)
* The participant has adequate hematologic function
* The participant must have adequate coagulation function
* If the participant has received prior anthracycline therapy as part of his or her first-line regimen, the participant is able to engage in ordinary physical activity without significant fatigue or dyspnea (equivalent to New York Heart Association Class I function)
* Because the teratogenicity of ramucirumab is not known, the participant, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods)
* Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment

Exclusion Criteria:

* The participant has documented and/or symptomatic brain or leptomeningeal metastases
* The participant has experienced any Grade 3 to 4 gastrointestinal (GI) bleeding within 3 months prior to enrollment
* The participant has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the treating physician
* The participant has ongoing or active psychiatric illness or social situation that would limit compliance with treatment
* The participant has uncontrolled or poorly controlled hypertension [>160 milliliter of mercury (mmHg) systolic or >100 mmHg diastolic for >4 weeks] despite standard medical management
* The participant has a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment
* The participant has received chemotherapy, radiotherapy, immunotherapy, or targeted therapy for gastric cancer within 2 weeks prior to enrollment
* The participant has received any investigational therapy within 30 days prior to enrollment
* The participant has undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment
* The participant has received prior therapy with an agent that directly inhibits vascular endothelial growth factor (VEGF) (including bevacizumab), or vascular endothelial growth factor receptor-2 (VEGFR-2) activity, or any antiangiogenic agent
* The participant is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs; including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted
* The participant has elective or planned major surgery to be performed during the course of the clinical trial
* The participant has a known allergy to any of the treatment components
* The participant is pregnant or breastfeeding
* The participant is known to be positive for infection with the human immunodeficiency virus (HIV)
* The participant has known alcohol or drug dependency
* The participant has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer, other noninvasive carcinoma, or in situ neoplasm
* The participant has a known hypersensitivity to ramucirumab or any of the excipients
* The patient may not have received more than 1 prior therapy in the metastatic setting.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (42):
- Austria (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Steyr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zams
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friedrichshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaiserslautern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mönchengladbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolfsburg
- Greece (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marousi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neo Faliro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- South Korea (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheong Ju-City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chuncheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deagu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gangnam-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gangwon Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guri-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyeonggi-do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonbuk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jongno-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Namdong-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seowon-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Suwon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ulsan